CLINICAL TRIAL: NCT00806247
Title: A Randomized, Double-Blind, Parallel-Arm, Placebo and Active Controlled Dose-Ranging Study of the Efficacy and Safety of Multiple Doses of CG5503 (Tapentadol) IR for Postoperative Pain Following Bunionectomy Surgery
Brief Title: A Randomized, Double-Blind, Parallel-Arm, Placebo and Active Controlled Dose-Ranging Study of the Efficacy and Safety of Multiple Doses of Tapentadol IR for Postoperative Pain Following Bunionectomy Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004189
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Pain; Postoperative Pain
Keywords: Tapentadol; Bunionectomy; Analgesia; Acute pain; Postsurgical pain
MeSH Terms: conditions — Pain; Pain, Postoperative; Agnosia; Acute Pain | interventions — Tapentadol

INTERVENTIONS:
Drug: tapentadol HCl

SUMMARY:
This study was to evaluate the efficacy and safety of dosing regimens of tapentadol HCl immediate release capsules for the treatment of postoperative pain over a period of 12 hours on the first day following a bunionectomy in men and women.

DETAILED DESCRIPTION:
Tapentadol hydrochloride is a centrally active analgesic (antinociceptive) compound. This was a multicenter, randomized, double-blind, parallel-group, placebo- and active-controlled dose study in men and nonpregnant, nonlactating women. The patients were at least 18 and no more than 75 years of age and experienced moderate to severe pain within 9 hours after removal of postoperative analgesia. The surgery was a standardized first metatarsal bunionectomy. Treatment of postsurgical pain after the 9 hr period was with either placebo, tapentadol, or oxycodone using various dosing regimens. The primary objective of this study was to evaluate the efficacy and safety of these treatments on total pain relief and total change in pain intensity over 12 hours and reporting of adverse events, laboratory values, vital signs, and ECGs. Secondary objectives included evaluation of several other pain measures, and drug pharmacokinetics and pharmacodynamics. Six patient treatment groups received study medication orally at 0, 4, and 8 hours with one of the following dosing regimens: 1) placebo, placebo, and placebo, 2) 93 mg, 93 mg, and 93 mg tapentadol IR, 3) 140 mg, 140 mg, and 140 mg tapentadol IR, 4) 140 mg, 70 mg, and 70 mg tapentadol IR, 5) 186 mg, 93 mg, and 93 mg tapentadol IR, and 6) 10 mg, 10 mg, and 10 mg oxycodone IR.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe pain intensity within 9 hours of the discontinuation of the popliteal block, and permitted supplemental systemic analgesics, if taken, during the postoperative surgical period
* Moderate to severe categorical pain intensity and a pain intensity VAS = 40 mm

Exclusion Criteria:

* Randomization less than 10 hours after initiation of the standardized first metatarsal bunionectomy
* History of seizure (including febrile seizure), or loss of consciousness due to head trauma
* Use of antiparkinsonian drugs, neuroleptics, anticonvulsants, monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants (TCAs), SSRIs, and SNRIs at any time within 30 days of surgery and throughout the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2005-01; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Primary objective was that at least 1 of the treatment regimens with tapentadol IR was superior to placebo as measured by the sum of total pain relief and sum of pain intensity difference over 12 hours (SPRID12) on the first day after a bunionectomy.

SECONDARY OUTCOMES:
Secondary objectives included evaluation of several additional pain measures, tolerability to treatments, and drug pharmacokinetics and pharmacodynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Randomized, Double-Blind, Parallel-Arm, Placebo and Active Controlled Dose-Ranging Study of the Efficacy and Safety of Multiple Doses of CG5503 IR for Postoperative Pain Following Bunionectomy Surgery — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=562&filename=CR004189_CSR.pdf